CLINICAL TRIAL: NCT05544773
Title: Comparing Trauma Severity Scores Injury Severity Score "ISS", Rapid Emergency Medicine Score "REMS" and Kampala Trauma Score "KTS" in Polytrauma Patients for Survival Prediction and ICU Admission in Assiut and Suez Canal University Hospitals.
Brief Title: Comparing Trauma Severity Scores Injury Severity Score "ISS", Rapid Emergency Medicine Score "REMS" and Kampala Trauma Score "KTS"
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Nassar, Principal Investigator , Emergency Medicine Resident, Assiut University
Other Study IDs: ISS-REMS-KTS
Record Dates: First submitted 2022-09-11; First posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Polytrauma
MeSH Terms: conditions — Multiple Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Trauma is defined as a physical injury from an external source of sudden onset and severity, which require immediate medical attention.Despite improvements in trauma systems worldwide, trauma continues to be one of the leading causes of death and disability in all age groups, especially the young and middle age group.

For studying the outcomes of trauma, accurate and reliable methodological tools are required for appropriate scoring of severity and outcome prediction . Trauma scores were designed to facilitate the triage of patients in the ER (emergency room), and identify patients with Polytrauma with low chances of survival. Those scores were meant to organize and improve the quality of trauma care systems, and to assess resources allocation.3 12 In 1969, Researchers developed the Abbreviated Injury Scale (AIS) to grade the severity of individual injuries. Attempting to summarize injury severity in patients with multiple traumas with a single number is almost difficult; therefore, multiple alternative scoring systems were proposed afterwards, each with its own problems and limitations.

More than 50 scoring systems have been published for the classification of trauma patients in the field, emergency room, and intensive care settings. There are three main groups of trauma scores: (a) Anatomical, (b) Physiological, (c) Combined scores. Anatomical scores describe all the injuries recorded by clinical examination, imaging, surgery or autopsy and measure lesion severity. Physiological scores describe changes happened due to the trauma, and translated by changes in vital signs and consciousness. Scores that include both anatomical and physiological criteria (mixed scores) are more useful for patient prognosis

DETAILED DESCRIPTION:
Trauma is defined as a physical injury from an external source of sudden onset and severity, which require immediate medical attention.Despite improvements in trauma systems worldwide, trauma continues to be one of the leading causes of death and disability in all age groups, especially the young and middle age group.

Approximately 5.8 million people die each year due to trauma related injuries, representing 8% of the worldwide mortality.Polytrauma is a short verbal equivalent commonly used for severely injured patients usually with associated injury (i.e. two or more severe injuries in at least two different areas of the body), less often with a multiple injury (i.e. two or more severe injuries in one body area).

Polytrauma patients usually have a much higher risk of mortalities and disabilities than the risk of expected mortalities in individual injuries patients. Even though polytrauma can occur due to different causes such as road traffic accidents, fall from heights, bullet injuries, suicide and homicide7.Yet the leading cause of traumatic related causes of death worldwide is road traffic accidents.8 Egypt, in particular, has experienced an alarming increase in the burden of traumatic injuries. According to the World Health Organization In 2015 Egypt has one of the highest rates of road accidents worldwide, with more than 12,000 fatalities each year, one of the highest among EMR countries. Although 90% of world's road trauma related fatalities occur in low- and middle-income countries, Injury prevention and trauma care programs in these countries have remained deficient.

For studying the outcomes of trauma, accurate and reliable methodological tools are required for appropriate scoring of severity and outcome prediction . Trauma scores were designed to facilitate the triage of patients in the ER (emergency room), and identify patients with Polytrauma with low chances of survival. Those scores were meant to organize and improve the quality of trauma care systems, and to assess resources allocation. In 1969, Researchers developed the Abbreviated Injury Scale (AIS) to grade the severity of individual injuries. Attempting to summarize injury severity in patients with multiple traumas with a single number is almost difficult; therefore, multiple alternative scoring systems were proposed afterwards, each with its own problems and limitations.

More than 50 scoring systems have been published for the classification of trauma patients in the field, emergency room, and intensive care settings. There are three main groups of trauma scores: (a) Anatomical, (b) Physiological, (c) Combined scores.

Anatomical scores describe all the injuries recorded by clinical examination, imaging, surgery or autopsy and measure lesion severity. Physiological scores describe changes happened due to the trauma, and translated by changes in vital signs and consciousness. Scores that include both anatomical and physiological criteria (mixed scores) are more useful for patient prognosis

The three types of scores can be combined in different ways to obtain more accurate information from all the possible aspects141- Anatomical Scoring Systems: Abbreviated injury scale (AIS) - Injury severity score (ISS) -New injury severity score (NISS) -Organ injury scale (OIS) - Anatomic profile -International Classification of Diseases (ICD-9) Injury Severity Score (ICISS) 2- Physiological Scoring Systems: Revised trauma score - Glasgow coma score - APACHE scoring (Acute physiology and chronic health evaluation - (APACHE I, II, III) -Rapid Emergency Medicine Score (REMS)3- Combined Anatomical and Physiological Scoring Systems :Trauma and injury severity scores (TRISS) - A severity characterization of trauma (ASCOT)-Kampala Trauma Score (KTS)

What does each score mean? Injury Severity Score (ISS): The injury severity score (ISS) is an anatomical scoring system which provides an overall score for patients with multiple injuries. Each injury is assigned an abbreviated injury scale (AIS) score and allocated to one of six body regions. The highest AIS score of each body region is used. The three most severely injured body regions scores are squared and added together to produce the ISS score.

Rapid Emergency Medicine Score (REMS): Rapid Emergency Medicine Score (REMS) is a newly developed scoring system developed to overcome drawbacks of other scoring systems. It is a simplified version of the APACHE II that allows for rapid score calculation. The REMS is calculated based on the patient's Glasgow Coma Scale (GCS), respiratory rate (RR), oxygen saturation, mean arterial pressure (MAP), heart rate (HR), and age.

Kampala Trauma Score (KTS): A new severity score, Kampala Trauma Score (KTS), was introduced as an injury severity score in settings without advanced diagnostics. This is a simplified composite of the Revised Trauma Score (RTS) and the Injury Severity Score (ISS). The KTS has been validated for its ability to predict outcome in the Ugandan trauma registry.

ELIGIBILITY:
Inclusion Criteria:

* traumatic patients with multiple trauma
* Both genders "without intently selected certain gender" and had 18 years old or more.

Exclusion Criteria:

* Patients who are less than 18 years old.
* Patients with end stage chronic disease .
* Patients with localized individual trauma will be excluded from this study.
* Patients refusing study .

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: traumatic patients with multiple trauma of both genders "without intently selected certain gender" and had 18 years old or more.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30 days
  Mortality "death" during the 30 day follow-up

SECONDARY OUTCOMES:
Hospital admission | Day 0
  Admission to hospital from the Emergency Department
Intensive Care Unit admission | Day 0
  Admission to the Intensive Care Unit or High Dependency Unit from the Emergency Department
Readmission in the Emergency Department | Hour 72, Day 30
  Re-visits to the Emergency Department after the index-visit.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lendrum RA, Lockey DJ. Trauma system development. Anaesthesia. 2013 Jan;68 Suppl 1:30-9. doi: 10.1111/anae.12049. PMID 23210554
- [Background] UF Health U of FH. Traumatic Injury. Published October 12, 2016. Accessed August 20, 2022. https://ufhealth.org/traumatic-injury
- [Background] Cernea D, Novac M, Dragoescu PO, Stanculescu A, Duca L, Al-Enezy AA, Dragoescu NA. Polytrauma and Multiple Severity Scores. Curr Health Sci J. 2014 Oct-Dec;40(4):244-8. doi: 10.12865/CHSJ.40.04.02. Epub 2014 Dec 14. PMID 26793320
- [Background] World Health Organization. Injuries and violence. Published March 19, 2021. Accessed August 20, 2022. https://www.who.int/news-room/fact-sheets/detail/injuries-and-violence
- [Background] Rau CS, Wu SC, Kuo PJ, Chen YC, Chien PC, Hsieh HY, Hsieh CH. Polytrauma Defined by the New Berlin Definition: A Validation Test Based on Propensity-Score Matching Approach. Int J Environ Res Public Health. 2017 Sep 11;14(9):1045. doi: 10.3390/ijerph14091045. PMID 28891977
- [Background] Marsden NJ, Tuma F. Polytraumatized Patient. 2023 Jul 3. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK554426/ PMID 32119313
- [Background] Bikbov B, Perico N, Remuzzi G. Mortality landscape in the global burden of diseases, injuries and risk factors study. Eur J Intern Med. 2014 Jan;25(1):1-5. doi: 10.1016/j.ejim.2013.09.002. Epub 2013 Sep 29. PMID 24084027
- [Background] The Global Road Safety Facility (GRSF), World Health Organization. Egypt's Road Safety Country Profile. Published 2016. Accessed August 20, 2022. https://www.roadsafetyfacility.org/country/egypt
- [Background] Elachi IC, Yongu WT, Odoyoh OO, Mue DD, Ogwuche EI, Ahachi CN. An epidemiological study of the burden of trauma in Makurdi, Nigeria. Int J Crit Illn Inj Sci. 2015 Apr-Jun;5(2):99-102. doi: 10.4103/2229-5151.158404. PMID 26157653
- [Background] Guzzo JL, Bochicchio GV, Napolitano LM, Malone DL, Meyer W, Scalea TM. Prediction of outcomes in trauma: anatomic or physiologic parameters? J Am Coll Surg. 2005 Dec;201(6):891-7. doi: 10.1016/j.jamcollsurg.2005.07.013. Epub 2005 Oct 13. PMID 16310692
- [Background] Knaus WA, Draper EA, Wagner DP, Zimmerman JE. APACHE II: a severity of disease classification system. Crit Care Med. 1985 Oct;13(10):818-29. PMID 3928249
- [Background] Le Gall JR. The use of severity scores in the intensive care unit. Intensive Care Med. 2005 Dec;31(12):1618-23. doi: 10.1007/s00134-005-2825-8. Epub 2005 Oct 22. No abstract available. PMID 16244878
- [Background] Beuran M, Negoi I, Paun S, Runcanu A, Gaspar B, Vartic M. [Trauma scores: a review of the literature]. Chirurgia (Bucur). 2012 May-Jun;107(3):291-7. Romanian. PMID 22844826
- [Background] Javali RH, Krishnamoorthy, Patil A, Srinivasarangan M, Suraj, Sriharsha. Comparison of Injury Severity Score, New Injury Severity Score, Revised Trauma Score and Trauma and Injury Severity Score for Mortality Prediction in Elderly Trauma Patients. Indian J Crit Care Med. 2019 Feb;23(2):73-77. doi: 10.5005/jp-journals-10071-23120. PMID 31086450
- [Background] Baker SP, O'Neill B, Haddon W Jr, Long WB. The injury severity score: a method for describing patients with multiple injuries and evaluating emergency care. J Trauma. 1974 Mar;14(3):187-96. No abstract available. PMID 4814394
- [Background] Olsson T, Terent A, Lind L. Rapid Emergency Medicine score: a new prognostic tool for in-hospital mortality in nonsurgical emergency department patients. J Intern Med. 2004 May;255(5):579-87. doi: 10.1111/j.1365-2796.2004.01321.x. PMID 15078500
- [Background] Kobusingye OC, Lett RR. Hospital-based trauma registries in Uganda. J Trauma. 2000 Mar;48(3):498-502. doi: 10.1097/00005373-200003000-00022. PMID 10744292
- [Background] MacLeod JBA, Kobusingye O, Frost C, Lett R, Kirya F, Shulman C. A Comparison of the Kampala Trauma Score (KTS) with the Revised Trauma Score (RTS), Injury Severity Score (ISS) and the TRISS Method in a Ugandan Trauma Registry. European Journal of Trauma. 2003;29(6):392-398. doi:10.1007/s00068-003-1277-5
- Available data/document: Study Protocol — https://drive.google.com/file/d/1gKwThkhpbD7eQxFYL4CkTEhzWtcLS1jZ/view?usp=sharing